CLINICAL TRIAL: NCT06028880
Title: Affirmative Mindfulness, Acceptance, and Compassion-based Group Intervention for Sexual Minorities (Free2Be): A Pilot Study
Brief Title: Affirmative Mindfulness, Acceptance, and Compassion-based Intervention for SM
Acronym: Free2Be
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Daniel Seabra, Daniel Seabra (Principal Investigator), University of Coimbra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Free2Be_intervention_SM; SFRH/BD/143437/2019 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Minority Stress
Keywords: Affirmative group intervention; Sexual Minorities; mindfulness; acceptance; compassion; stress; minority stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 1 pre-session + 12 sessions
  Interventions: Behavioral: Free2Be

INTERVENTIONS:
Behavioral: Free2Be — Free2Be is a manualized 13-week face-to-face group intervention for SM individuals with one pre-session and plus 12 intervention sessions. The themes of each session are: Human nature & Relation with suffering (S1), Emotional regulation & Multiple selves (S2), Creative hopelessness & Values (S3), Compassionate attention (S4), Compassionate acceptance (S5), Self-criticism; Compassion & Flows of compassion (S6), Compassionate imagination; Compassionate self (S7), Early experiences; Stigma and shame; & Compassionate cognitive desfusion (S8), Compassionate thinking (S9), Difficult emotions: Shame & Anger (S10), Coming out & Compassionate behaviour (assertiveness) (S11), Positive emotions & Preparing for the future (S2).

SUMMARY:
The goal of this pilot clinical trial is to explore the effectiveness of Free2Be group intervention for sexual minorities. The main questions it aims to answer are:

* Is it Free2Be effective in the decrease of stress?
* Are mindfulness, acceptance, and self-compassion responsible for changes in psychological symptoms?

Participants will receive an affirmative mindfulness, acceptance, and self-compassion-based face-to-face group intervention with 13 weekly sessions (Free2Be).

DETAILED DESCRIPTION:
Sexual Minorized (SM) individuals include several self-identified nonheterosexual sexual orientations. This population face uncountable forms of discrimination stemming from social stigma. Unsurprisingly, levels of psychopathology are poorer in SM individuals when compared to heterosexual individuals, The Minority Stress Model describes stress processes that help to explain this disparity, for example, expectations of rejection and internalized stigma. Beyond the specific minority-related processes, general maladaptive psychological processes also contribute to the elevated risk of psychopathology in this population (Psychological Mediation Framework), for example, self-criticism. Additionally, shame and fears of compassion seem to affect the mental health in this population.

When SM individuals try to access mental health care, they find inappropriate and discriminatory services with professionals without specific training on sexuality-related themes. Affirmative interventions are wide approaches with a positive and respectful perspective about sexual orientations, recognizing different identities as representations of human diversity. This approach identifies negative consequences in mental health as consequences of stress related to heterosexism, discrimination and violence against SM individuals.

Previous studies reinforcing the relevance of mindfulness, acceptance, and self-compassion as positive psychological processes for SM individuals. Free2Be was the first affirmative intervention based on mindfulness, acceptance, and compassion techniques for SM individuals, and is a manualized 13 weeks, face-to-face group intervention. The feasibility results highlighted the acceptability of this intervention, suggested some changes in the intervention content, and concluded about the viability of a pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Majority (> 18 years old)
* Nonheterosexual self-identified
* Being Portuguese
* Perfectly understanding of Portuguese oral and written language
* Gave informed and free consent

Exclusion Criteria:

* Currently receiving individual or group psychotherapy
* Major Depressive Disorder - severe specifier
* Hypo/maniac Episode - without full remission
* Psychosis Characteristics in the last two months
* Social impairment from Substance Use Disorder
* High suicide risk (according to the Suicide Risk Index).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Stress symptoms assessed by DASS-21 | 6 months (from Baseline to 3-months follow-up)
  The subscale Stress symptoms of the self-report Depression Anxiety Stress Scales (Lovibond & Lovibond, 1995; Pais-Ribeiro et al., 2004) has 7 items that assess difficulties in relaxing, nervous excitement, agitation, exaggerated reactions, and impatience.

SECONDARY OUTCOMES:
Mindfulness assessed by CompACT-18 | 6 months (from Baseline to 3-months follow-up)
  The subscale Behavioural awareness of the self-report Comprehensive assessment of Acceptance and Commitment Therapy processes - 18 Items (CompACT-18; Francis et al., 2016; Trindade et al., 2021) has 5 items that assess mindful attention to the present moment.
Acceptance assessed by CompACT-18 | 6 months (from Baseline to 3-months follow-up)
  The subscale Openness to experience of the self-report Comprehensive assessment of Acceptance and Commitment Therapy processes - 18 Items (CompACT-18; Francis et al., 2016; Trindade et al., 2021) has 5 items that assess willingness to allow internal experiences without efforts to change it.
Self-compassion assessed by CMAS | 6 months (from Baseline to 3-months follow-up)
  The Self-compassion scale of the self-report Compassion Motivation and Action Scales (CMAS; Steindl et al., 2021; Matos et al., 2023) has 18 items that assess the intent to be self-compassionate, distress tolerance during own suffering, and behaviours to alleviate this suffering.
Stigma consciousness assessed by SCQ-PT | 6 months (from Baseline to 3-months follow-up)
  The self-report Stigma Consciousness Questionnaire (SCQ-PT; Pinel, 1999; Seabra, Gato, et al., 2023) has 10 items that assess the extent to which sexual minority individuals focus on feel self-conscious about their stereotyped status.
Internalized stigma assessed by LGBIS | 6 months (from Baseline to 3-months follow-up)
  The subscale Identity dissatisfaction of the self-report Lesbian, Gay, Bisexual Identity Scale (LGBIS; Mohr & Kendra, 2011; Oliveira et al., 2012) has 6 items that assess internalized stigma.
Shame assessed by SMEISS | 6 months (from Baseline to 3-months follow-up)
  The Sexual Minority External and Internal Shame Scale (Manão et al., 2023) has 8 items that assess shame related to sexual orientation.
Self-Criticism assessed by FSCRS | 6 months (from Baseline to 3-months follow-up)
  The composite measure of Inadequate self and Hated self of the self-report Forms of Self-criticizing/Attacking and Self-reassuring Scale (FSCRS; Gilbert et al., 2004; Castilho et al., 2015) has 14 items that assess the experience of inadequacy and self-dislike when failures and setbacks occur. The use of this composite measure is very common in the assessment of self-criticism. Recent years research in non-clinical samples has favoured a unique global factor of self-criticism considering Inadequate self and Hated self together (Halamová et al., 2019).
Fears of compassion for other assessed by FCS | 6 months (from Baseline to 3-months follow-up)
  The subscale Fear of compassion to others of the self-report Fears of Compassion Scale (FCS; Gilbert et al., 2011; Simões, 2012) has 10 items that assess fears, blocks, and resistances to giving compassion to others.
Fears of compassion from other assessed by FCS | 6 months (from Baseline to 3-months follow-up)
  The subscale Fear of compassion from others of the self-report Fears of Compassion Scale (FCS; Gilbert et al., 2011; Simões, 2012) has 13 items that assess fears, blocks, and resistances to receive compassion.
Fears of self-compassion assessed by FCS | 6 months (from Baseline to 3-months follow-up)
  The subscale Fear for compassion for self of the self-report Fears of Compassion Scale (FCS; Gilbert et al., 2011; Simões, 2012) has 15 items that assess one's fears, blocks, and resistances to self-compassion.
Anxiety symptoms assessed by DASS-21 | 6 months (from Baseline to 3-months follow-up)
  The subscale Anxiety symptoms of the self-report Depression Anxiety Stress Scales (Lovibond & Lovibond, 1995; Pais-Ribeiro et al., 2004) has 7 items that assess physical arousal symptoms, panic attacks, and fear.
Depressive symptoms assessed by DASS-21 | 6 months (from Baseline to 3-months follow-up)
  The subscale Depression symptoms of the self-report Depression Anxiety Stress Scales (Lovibond & Lovibond, 1995; Pais-Ribeiro et al., 2004) has 7 items that assess symptoms usually associated with negative mood.
Social anxiety symptoms assessed by SIAS | 6 months (from Baseline to 3-months follow-up)
  The self-report Social Interaction Anxiety Scale (SIAS; Mattick & Clarke, 1998; Pinto-Gouveia & Salvador, 2001) has 19 items that assess fears of general social interaction.
Positive affect (drive system) assessed by ASCAS | 6 months (from Baseline to 3-months follow-up)
  The composite measure of Activated positive affect and Relaxed positive affect of the self-report Activation and Safe/Content Affect Scale (ASCAS; Gilbert et al., 2008; Pinto-Gouveia et al., 2008) has 14 items that assess the experience of positive affect associated to resource acquisitions and achievements. This composite measure aligns with theorical affect regulation systems (Gilbert, 2010).
Positive affect (soothing system) assessed by ASCAS | 6 months (from Baseline to 3-months follow-up)
  The subscale Safe/content positive affect of the self-report Activation and Safe/Content Affect Scale (ASCAS; Gilbert et al., 2008; Pinto-Gouveia et al., 2008) has 4 items that assess the experience of positive affect associated to safeness, caring, and contentment.
Negative affect (threat system) assessed by PANAS | 6 months (from Baseline to 3-months follow-up)
  The subscale Negative affect of the self-report Positive and Negative Affect Schedule (PANAS; Watson, Clark & Tellegen, 1988; Galinha & Pais-Ribeiro, 2005) has 10 items that assess the experience of positive affect associated to detection and protection.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Seabra, Principal Investigator — University of Coimbra
Locations (2):
- Portugal (2):
  - Faculty of Psychology and Educational Science, Coimbra
  - Serviços De Acção Social Da Universidade De Coimbra, Coimbra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pachankis JE. Uncovering Clinical Principles and Techniques to Address Minority Stress, Mental Health, and Related Health Risks Among Gay and Bisexual Men. Clin Psychol (New York). 2014 Dec;21(4):313-330. doi: 10.1111/cpsp.12078. PMID 25554721
- [Background] Helminen EC, Ducar DM, Scheer JR, Parke KL, Morton ML, Felver JC. Self-Compassion, Minority Stress, and Mental Health in Sexual and Gender Minority Populations: A Meta-Analysis and Systematic Review. Clin Psychol (New York). 2023 Mar;30(1):26-39. doi: 10.1037/cps0000104. Epub 2022 Nov 28. PMID 37197599
- [Background] Fowler JA, Buckley L, Muir M, Viskovich S, Paradisis C, Zanganeh P, Dean JA. Digital mental health interventions: A narrative review of what is important from the perspective of LGBTQIA+ people. J Clin Psychol. 2023 Nov;79(11):2685-2713. doi: 10.1002/jclp.23571. Epub 2023 Aug 2. PMID 37528773
- [Background] Meyer IH. Prejudice, social stress, and mental health in lesbian, gay, and bisexual populations: conceptual issues and research evidence. Psychol Bull. 2003 Sep;129(5):674-697. doi: 10.1037/0033-2909.129.5.674. PMID 12956539